CLINICAL TRIAL: NCT03368404
Title: A Study to Evaluate the Performance and Safety of CBL-102 Versus Vismed® Multi Eye Drops in the Management of Dry Eye
Acronym: RESTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire Chauvin (Industry)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBL-2017-01; 2017-A01099-44 (Other: ANSM Registry Office RCB - France)
Record Dates: First submitted 2017-11-28; First posted 2017-12-11 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye
Keywords: dry eye, tear substitute, ocular lubricant
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBL-102 eye drops (Experimental): CE marked medical device, tear substitute containing 0.24% hyaluronic acid salt, carbomer and medium chain triglycerides, presented in 10 mL bottles
  Interventions: Device: CBL-102 eye drops
- Vismed Multi eye drops (Active Comparator): CE marked medical device, tear substitute containing 0.18% sodium hyaluronate, presented in 10 mL bottles
  Interventions: Device: Vismed Multi eye drops

INTERVENTIONS:
Device: CBL-102 eye drops — CBL-102 eye drops, 3 to 6 times per day for 3 months
  Arms: CBL-102 eye drops
Device: Vismed Multi eye drops — Vismed Multi eye drops, 3 to 6 times per day for 3 months
  Arms: Vismed Multi eye drops

SUMMARY:
The primary objectives of this investigation were to show that the performance of CBL-102 Eye Drops is non-inferior to that of Vismed® Multi eye drops in subjects with moderate to severe keratoconjunctivitis sicca after 28 days, and to assess the safety of CBL-102 Eye Drops during a 90-day period with treatment administered 3 to 6 times per day.

DETAILED DESCRIPTION:
This was a multicenter, randomized, parallel group, investigator-masked, non-inferiority study. Approximately 84 subjects were planned to be randomized in a 1:1 ratio.

The primary performance endpoint was the mean change from baseline (CFB) in the study eye at Day 28 in the Ocular surface fluorescein staining score as assessed by the Oxford Scheme.

Following a screening visit (Visit 1) and a 2-week washout with povidone 2% artificial tear (ART), participants were randomized on Day 0 (Visit 2) with follow-up visits on Day 28 ±3 (Visit 4) and Day 90 ±10 (Visit 5). A telephone assessment took place on Day 7 ±1 ('Visit 3') for safety and compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 and ability to read, understand, and provide written voluntary informed consent on the Ethics Committee approved Informed Consent Form
2. Ability and willingness to comply with all treatment and follow-up and study procedures
3. Use of tear substitutes for at least 2.5 months prior to inclusion, and agreement to use multidose preservative-free ART (Aqualarm® U.P. povidone 2% eye drops in 10 mL bottles) up to 6 times a day for at least 2 weeks immediately prior to randomization
4. Symptom score ≥ 1 for at least 2 out of the 7 following symptoms (rated 0 to 4): sensation of dryness, foreign body, burning, stinging, itching, blurred vision, sensitivity to light
5. At least 1 eye with the following signs of keratoconjunctivitis sicca :

   * Tear break-up time of 10 sec (mean of 3 measurements) at both screening visit and inclusion visit
   * Total ocular surface staining score ≥ 4 and ≤ 9 at both screening visit and inclusion visit. This assessment combines corneal, nasal and temporal bulbar conjunctival fluorescein staining, each graded 0-5 according to the Oxford Scheme
6. A decimal visual acuity with habitual correction equal to or better than 0.1 (Monoyer chart) in both eyes
7. No systemic treatment or who had received stable systemic treatment (unchanged for 1 month or longer)
8. Female subjects had to be into 1 of the following categories:

   * Post-menopausal
   * Surgically sterile
   * Using birth control method throughout the duration of the study
9. Female of childbearing potential needed a negative urine pregnancy test result at screening

Exclusion Criteria:

1. Severe blepharitis
2. Severe ocular dryness accompanied by 1 of the following:

   * Lid abnormality
   * Corneal disease
   * Ocular surface metaplasia
   * Filamentary keratitis
   * Corneal neovascularization
3. Use of contact lenses at inclusion or within 90 days prior to study start
4. History of ocular surgery, including laser surgery, in either eye within 180 days prior to study start
5. History of ocular trauma, non-dry eye ocular inflammation, or ocular infection within 90 days prior to study start
6. History of ocular allergic disease or ocular herpes within 1 year prior to study start
7. History of any inflammatory ulcerative keratitis, recurrent corneal erosion, or uveitis
8. Known hypersensitivity or contraindications to any of the ingredients in the test or comparator products or ART
9. Initiation of, or changes to, concomitant medication that could affect dry eye within 30 days prior to Visit 1 (Screening) or with planned initiation or changes of such medications during the study
10. Ocular therapy (either eye) with any ophthalmic medication, except tear substitutes, within 2 weeks prior to study start
11. Expected use of ocular therapy during the study
12. Use of topical ocular steroidal or non-steroidal anti-inflammatory medication within 30 days prior to study start
13. Expected use of ocular therapy with immunosuppressants during the study or use of ocular immunosuppressants within 90 days prior to study start
14. Use of occlusion therapy with non-resorbable lacrimal or punctum plugs within 90 days prior to study start or use of resorbable plugs
15. Use or planned use of therapy such as LipiFlow® or BlephEx®
16. Breastfeeding females
17. Participation in any drug or device clinical investigation within 30 days prior to entry into study and/or during the period of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Labetoulle, M.D Ph.D, Principal Investigator — Hôpital Kremlin-Bicêtre
Locations (1):
- Hôpital Kremlin-Bicêtre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 16 sites in France
Pre-assignment Details: 92 enrolled participants underwent a washout period of 2 weeks with povidone 2% eye drops in both eyes. Following completion of the washout period, 87 participants met inclusion criteria and were randomized either to CBL-202 or Vismed Multi treatment group. Both eyes of each participant were treated with assigned eye drops.
Groups:
- CBL-102 Eye Drops: Participants received CBL-102 Eye Drops, 3 to 6 times daily for 3 months in both eyes.
  CBL-102 Eye Drops: CE-marked medical device, tear substitute with 0.24% sodium hyaluronate, carbomer and triglycerides
- Vismed® Multi Eye Drops: Participants received Vismed® Multi eye drops, 3 to 6 times daily for 3 months in both eyes.
  Vismed® Multi: CE-marked medical device, tear substitute with 0.18% sodium hyaluronate
Period: Overall Study
Arm/Group | CBL-102 Eye Drops | Vismed® Multi Eye Drops
Started | 48 (One participant never took the assigned product and withdrew consent.) | 39 (One participant did not have the Day 28 performance assessments and was withdrawn from the Intention-to-treat population according to the protocol. The participant was included in the Safety population.)
Safety Population | 47 | 39
Intention-to-treat- Population | 47 | 38
Per Protocol Population Day 28 | 45 | 34
Per Protocol Population Day 90 | 44 | 33
Completed | 45 | 37
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data were only collected for Intention-to-treat population. Intention-to-treat-population: all participants with treatment and a post-baseline assessment Each Baseline Participant contributed one study eye.
Groups:
- Total: Total of all reporting groups
Arm/Group | CBL-102 Eye Drops | Vismed® Multi Eye Drops | Total
Number analyzed (Participants) | 47 | 38 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (14.3) | 64.8 (14.7) | 63.6 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 27 | 59
  Male | 15 | 11 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 47 | 38 | 85
Ocular surface fluorescein staining [Mean (Standard Deviation); unit: units on a scale] — The Ocular Surface Fluorescein Score (OSFS) was scored according to scale (Oxford Scheme) with total score ranging from a minimum of 0 (best outcome) to a maximum of 15 (worst outcome).
  The total OSFS total score is the sum of 3 sub-scores (corneal, nasal and temporal regions).
  Each sub-score ranges from a minimum of 0 (best outcome) to a maximum of 5 (worst outcome).
  units on a scale | 5.7 (1.2) | 5.9 (1.3) | 5.8 (1.3)
Corneal fluorescein staining score [Mean (Standard Deviation); unit: units on a scale] — The Corneal fluorescein staining score was measured according to a scale (Oxford Scheme) ranging from 0 (best outcome) to 5 (worst outcome).
  units on a scale | 1.9 (0.8) | 1.9 (0.9) | 1.9 (0.8)
Nasal conjunctival fluorescein staining score [Mean (Standard Deviation); unit: units on a scale] — The Nasal fluorescein staining score was measured according to a scale (Oxford Scheme) ranging from 0 (best outcome) to 5 (worst outcome).
  units on a scale | 1.9 (0.6) | 1.9 (0.7) | 1.9 (0.6)
Temporal conjunctival fluorescein staining score [Mean (Standard Deviation); unit: units on a scale] — The Temporal fluorescein staining score was measured according to a scale (Oxford Scheme) ranging from 0 (best outcome) to 5 (worst outcome).
  units on a scale | 1.9 (0.6) | 2.1 (0.6) | 2.0 (0.6)
Global dry eye symptoms score [Mean (Standard Deviation); unit: units on a scale] — The Global dry eye symptom score was the sum score (scale 0-28) of dry eye symptoms assessing 7 items: sensation of dryness, foreign body, burning, stinging, itching, blurred vision, sensitivity to light), each graded individually from 0 (absence) to 4 (severe and/or disabling and constant).
  units on a scale | 11.0 (3.8) | 9.0 (3.8) | 10.1 (3.9)
Ocular surface disease-Quality of life (OSD-QoL®) [Mean (Standard Deviation); unit: units on a scale] — The OSD-QoL® questionnaire is a validated instrument for measuring dry eye severity and impairment. It includes 28 items divided into 7 dimensions: Daily activities, Difficulties with work and handicap, Giving up makeup, Acknowledgement of the disease, Acceptance of the disease, Fear for the future, and Emotional well-being.
  A Global Question: "How do you feel when considering your eye problems?" (included in the Fear for the future dimension) is also evaluated separately. The converted score for each dimension ranges from 0-100, with a higher score reflecting a better quality of life. Population: Some of the Quality-of-Life questionnaires could not be analyzed due to incomplete data.
  Giving up makeup dimension was only completed by women.
  units on a scale
    Daily activities: number analyzed (Participants) | 44 | 36 | 80
    Daily activities | 65.9 (19.6) | 64.7 (24.5) | 65.4 (21.8)
    Difficulties with work and handicap: number analyzed (Participants) | 37 | 30 | 67
    Difficulties with work and handicap | 75.1 (17.7) | 74.9 (22.4) | 75.0 (19.8)
    Giving up makeup: number analyzed (Participants) | 25 | 24 | 49
    Giving up makeup | 63.0 (33.2) | 54.2 (35.1) | 58.7 (34.1)
    Acknowledgement of the disease: number analyzed (Participants) | 44 | 36 | 80
    Acknowledgement of the disease | 34.9 (19.9) | 31.3 (19.2) | 33.3 (19.6)
    Acceptance of the disease: number analyzed (Participants) | 44 | 36 | 80
    Acceptance of the disease | 76.7 (24.4) | 61.8 (35.6) | 70.0 (30.7)
    Fear for the future: number analyzed (Participants) | 43 | 36 | 79
    Fear for the future | 59.2 (16.9) | 55.1 (19.9) | 57.3 (18.3)
    Emotional well-being: number analyzed (Participants) | 44 | 35 | 79
    Emotional well-being | 82.7 (19.3) | 80.0 (20.6) | 81.5 (19.8)
    Global Question: number analyzed (Participants) | 44 | 36 | 80
    Global Question | 50.6 (19.8) | 50.0 (23.1) | 50.3 (21.2)
Tear film break-up time (TFBUT) [Mean (Standard Deviation); unit: seconds] — The Tear Film Break Up Time (TFBUT) is assessed after fluorescein instillation and is the time measured between the last blink and the first appearance of a dry spot or disruption of the tear film. The TFBUT was measured in tenths of seconds with a stopwatch provided to the sites. It was conducted 3 times and the mean was calculated.
  seconds | 5.9 (1.7) | 5.4 (1.9) | 5.7 (1.8)
Schirmer's test [Mean (Standard Deviation); unit: millimeters] — Tear fluid secretion was assessed by un-anaesthetised Schirmer's test in the study eye with graduated strips in millimetres.
  Schirmer paper test strips were carefully inserted over the lower eyelid margin. The strips were removed after 5 minutes and the amount of tear fluid secretion was read to the nearest mm from the graduated strip margin.
  millimeters | 7.2 (5.0) | 7.1 (4.8) | 7.1 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ocular Surface Fluorescein Staining Score at Day 28
Description: Mean change from baseline (CFB) in the study eye in Ocular Surface Fluorescein Staining (OSFS) scored according to the Oxford Scheme.
  The Oxford Scheme is a validated scale consisting of a series of panels labelled A to E in order of increasing severity. Grade 0 corresponds to panel A increasing to Grade 5 corresponding to more than Panel E, with punctate dots representing staining. The 3 regions, cornea, nasal and temporal bulbar conjunctiva are graded separately from 0 (best outcome) to 5 (worst outcome), with the Ocular Surface Fluorescein Score (OSFS) ranging from 0 (best outcome) to 15 (worst outcome). The OSFS is the sum score of the 3 sub-scores (corneal, nasal and temporal regions).
  The study eye was the eligible eye with the highest OSFS score at baseline, which needed to be ≥4 and ≤9 on the 15-grade Oxford Scheme. If both eyes were eligible and had the same OSFS score, the study eye was the right eye.
Time Frame: Baseline (Day 0), Visit 4 (Day 28)
Population: Per-protocol population: all randomized participants with at least one instillation and one post-baseline assessment without any major protocol deviation (defined as impacting the primary endpoint)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-102 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 45 | 34
score on a scale | -2.1 (0.2) | -1.5 (0.3)
Statistical Analysis 1: Comparison: CBL-102 Eye Drops vs Vismed® Multi Eye Drops; Test type: Non-Inferiority — A sample size of 33 evaluable patients per treatment group was calculated to provide at least 90% power to demonstrate non-inferiority of CBL-102 to Vismed Multi. Assumptions included a non-inferiority margin of 2 grades and a standard deviation of 2.5; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.34 to 0.13], Standard Error of Mean 0.4 — Treatment difference : CBL-102 - Vismed Multi

2. Secondary Outcome: Change From Baseline in Ocular Surface Fluorescein Staining Score at Day 90 (Visit 5)
Description: Mean change from baseline (CFB) in the study eye in Ocular Surface Fluorescein Staining (OSFS) scored according to the Oxford Scheme.
  The Oxford Scheme is a validated scale consisting of a series of panels labelled A to E in order of increasing severity. Grade 0 corresponds to panel A increasing to Grade 5 corresponding to more than Panel E, with punctate dots representing staining. The 3 regions, cornea, nasal and temporal bulbar conjunctiva are graded separately from 0 to 5, with the OSFS score ranging from 0 (best outcome) to 15 (worst outcome).
  The study eye was the eligible eye with the highest OSFS score at baseline, which needed to be ≥4 and ≤9 on the 15-grade Oxford Scheme. If both eyes were eligible and had the same OSFS score, the study eye was the right eye.
Time Frame: Baseline (Day 0), Visit 5 (Day 90)
Population: Two participants of per-protocol population, one in each group withdrew before Day 90 visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- CBL-102 Eye Drops: Participants received CBL-102 Eye Drops, 3 to 6 times daily for 3 months in both eyes.
  CBL-102 Eye Drops: CE-marked medical device, tear substitute wit 0.24% sodium hyaluronate, carbomer and triglycerides
- Vismed Multi Eye Drops: Participants received Vismed ® Multi eye drops, 3 to 6 times daily for 3 months in both eyes.
  Vismed ® Multi: CE marked medical device, tear substitute with 0.18% sodium hyaluronate
Arm/Group | CBL-102 Eye Drops | Vismed Multi Eye Drops
Number analyzed (Participants) | 44 | 33
score on a scale | -3.1 (0.3) | -2.3 (0.3)
Statistical Analysis 1: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Test type: Superiority; p = 0.0592, ANCOVA — Significance level of 0.05; Adjustment for baseline

3. Secondary Outcome: Change From Baseline in Corneal Fluorescein Staining Score at Day 28 (Visit 4) and at Day 90 (Visit 5)
Description: Mean change from baseline (CFB) in the study eye in Corneal Fluorescein Staining (OSFS) scored according to the Oxford Scheme.
  The Oxford Scheme is a validated scale consisting of a series of panels labelled A to E in order of increasing severity. Grade 0 corresponds to panel A increasing to Grade 5 corresponding to more than Panel E, with punctate dots representing staining. The Corneal Region is graded separately from 0 (best outcome) to 5 (worst outcome).
Time Frame: Baseline (Day 0), Visit 4 (Day 28) and Visit 5 (Day 90)
Population: Two participants of the per-protocol population, one in each group withdrew before the Day 90 visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-102 Eye Drops | Vismed Multi Eye Drops
Number analyzed (Participants) | 45 | 34
score on a scale
  CFB in Corneal Fluorescein Score at Day 28 (Visit 4) | -0.8 (0.1) | -0.6 (0.1)
  CFB in Corneal Fluorescein Score at Day 90 (Visit 5): number analyzed (Participants) | 44 | 33
  CFB in Corneal Fluorescein Score at Day 90 (Visit 5) | -1.0 (0.1) | -0.8 (0.1)
Statistical Analysis 1: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Test type: Superiority; p > 0.05, ANCOVA — Significance level of 0.05; Adjustment for baseline

4. Secondary Outcome: Change From Baseline in Nasal Conjunctival Fluorescein Staining Score at Day 28 (Visit 4) and at Day 90 (Visit 5)
Description: Mean change from baseline (CFB) in the study eye in Nasal Conjunctival Fluorescein Staining scored according to the Oxford Scheme.
  The Oxford Scheme is a validated scale consisting of a series of panels labelled A to E in order of increasing severity. Grade 0 corresponds to panel A increasing to Grade 5 corresponding to more than Panel E, with punctate dots representing staining. The Nasal conjunctival region is graded separately from 0 (best outcome) to 5 (worst outcome).
Time Frame: Baseline (Day 0), Visit 4 (Day 28) and Visit 5 (Day 90)
Population: Two participants of the per-protocol population, one in each group withdrew before Day 90 (Visit 5)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-102 Eye Drops | Vismed Multi Eye Drops
Number analyzed (Participants) | 45 | 34
score on a scale
  Change from Baseline in NAsal Conjunctival Fluorescein Staining Score at Day 28 (Visit 4) | -0.6 (0.1) | -0.4 (0.1)
  Change from Baseline in Nasal Conjunctival Fluorescein Staining Score at day 90 (Visit 5): number analyzed (Participants) | 44 | 33
  Change from Baseline in Nasal Conjunctival Fluorescein Staining Score at day 90 (Visit 5) | -0.9 (0.1) | -0.6 (0.2)
Statistical Analysis 1: Comparison: CBL-102 Eye Drops; Test type: Superiority; p > 0.05, ANCOVA — Significance level 0.05; Adjustment for baseline

5. Secondary Outcome: Change From Baseline in Temporal Conjunctival Fluorescein Staining Score at Day 28 (Visit 4) and at Day 90 (Visit 5)
Description: Mean change from baseline (CFB) in the study eye in Temporal Conjunctival Fluorescein Staining scored according to the Oxford Scheme.
  The Oxford Scheme is a validated scale consisting of a series of panels labelled A to E in order of increasing severity. Grade 0 corresponds to panel A increasing to Grade 5 corresponding to more than Panel E, with punctate dots representing staining. The Temporal Conjunctival region is graded separately from 0 (best outcome) to 5 (worst outcome).
Time Frame: Baseline (Day 0), Visit 4 (Day 28), Visit 5 (Day 90)
Population: Two participants of the per-protocol population, on in each group withdrew before Day 90 (Visit 5)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-102 Eye Drops | Vismed Multi Eye Drops
Number analyzed (Participants) | 45 | 34
score on a scale
  Change From Baseline in temporal Conjunctival Staining Score at Day 28 (Visit 4) | -0.8 (0.1) | -0.4 (0.1)
  Change From BAseline in Temporal Conjunctival Staining Score at Day 90 (Visit 5): number analyzed (Participants) | 44 | 33
  Change From BAseline in Temporal Conjunctival Staining Score at Day 90 (Visit 5) | -1.2 (0.1) | -0.9 (0.1)
Statistical Analysis 1: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Test type: Superiority; p > 0.05, ANCOVA — Significance level of 0.05; Adjustment for baseline

6. Secondary Outcome: Change From Baseline in Global Sum Score of Dry Eye Symptoms at Day 28 (Visit 4) and at Day 90 (Visit 5)
Description: The global sum score (scale 0-28) of dry eye symptoms assessed 7 items: sensation of dryness, foreign body, burning, stinging, itching, blurred vision, sensitivity to light, each graded from 0 (absent) to 4 (severe and/or disabling and constant).
Time Frame: Baseline (Day 0), Visit 4 (Day 28) and Visit 5 (Day 90)
Population: Two participants of the per-protocol population, one in each group withdrew before the Day 90 visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-102 Eye Drops | Vismed Multi Eye Drops
Number analyzed (Participants) | 45 | 34
score on a scale
  Change From Baseline in Global Sum Score of Dry Eye Symptoms at Day (Visit 4) | -3.9 (0.5) | -2.1 (0.5)
  Change From Baseline in Global Sum Score of Dry Eye Symptoms at Day 90 (Visit 5): number analyzed (Participants) | 44 | 33
  Change From Baseline in Global Sum Score of Dry Eye Symptoms at Day 90 (Visit 5) | -6.3 (0.5) | -3.9 (0.5)
Statistical Analysis 1: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Change from Baseline in Global Sum Score of Dry Eye Symptoms at Day 28 (Visit 4); Test type: Superiority; p = 0.0176, ANCOVA — Significance level 0.05
Statistical Analysis 2: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Change from Baseline in Global Sum Score of Dry Eye Symptoms at Day 90 (Visit 5); Test type: Superiority; p = 0.0010, ANCOVA — Significance level 0.05; Adjustment to baseline

7. Secondary Outcome: Change From Baseline in the Ocular Surface Disease-Quality of Life (OSD-QoL®) at Day 90 (Visit 5)
Description: The OSD-QoL® questionnaire is a validated instrument for measuring dry eye severity and impairment. It includes 28 items divided into 7 dimensions: Daily activities, Difficulties with work and handicap, Giving up makeup, Acknowledgement of the disease, Acceptance of the disease, Fear for the future, and Emotional well-being. A Global Question: "How do you feel when considering your eye problems?" (included in the Fear for the future dimension) is also evaluated separately. The converted score for each dimension ranges from 0 to 100, with a higher score reflecting a better quality of life.
Time Frame: Baseline (Day 0), Visit 5 (Day 90)
Population: Analysis population included participants in the per-protocol population with evaluable Questionnaire dimension or Global question on both Day 0 and Day 90.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-102 Eye Drops | Vismed Multi Eye Drops
Number analyzed (Participants) | 40 | 31
score on a scale
  Daily activities | 11.3 (1.9) | 4.8 (2.1)
  Difficulties with work and handicap: number analyzed (Participants) | 34 | 22
  Difficulties with work and handicap | 9.8 (1.5) | 1.6 (1.9)
  Giving up makeup: number analyzed (Participants) | 19 | 22
  Giving up makeup | 14.1 (3.9) | 7.1 (3.7)
  acknowledgement of the disease | 5.1 (2.7) | -3.3 (3.0)
  acceptance of the disease | 2.7 (3.4) | -1.8 (3.9)
  Fear for the future: number analyzed (Participants) | 39 | 31
  Fear for the future | 10.8 (2.1) | 4.6 (2.4)
  Emotional well-beig: number analyzed (Participants) | 39 | 30
  Emotional well-beig | 5.5 (2.0) | 4.4 (2.2)
  Global Question: number analyzed (Participants) | 40 | 30
  Global Question | 17.6 (2.4) | 9.5 (2.8)
Statistical Analysis 1: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Ocular Surface Disease-Quality of Life (OSD-QoL®) dimension: Daily Activities; Test type: Superiority; p = 0.0251, ANCOVA — Significance level 0.05; Adjustment for baseline
Statistical Analysis 2: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Ocular Surface Disease-Quality of Life (OSD-QoL®) dimension: Difficulties with work and handicap; Test type: Superiority; p = 0.0015, ANCOVA — Significance level of 0.05; Adjustment for baseline
Statistical Analysis 3: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Ocular Surface Disease-Quality if Life (OSD-QoL®) dimension: Giving up makeup; Test type: Superiority; p = 0.2024, ANCOVA — Significance level 0.05; Adjustment for baseline
Statistical Analysis 4: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Ocular Surface Disease-Quality if Life (OSD-QoL®) dimension: Acknowledgement of the Disease; Test type: Superiority; p = 0.0421, ANCOVA — Significance level 0.05; Adjustment for baseline
Statistical Analysis 5: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Ocular Surface Disease-Quality if Life (OSD-QoL®) dimension: Acceptance of the disease; Test type: Superiority; p = 0.3945, ANCOVA — Significance level 0.05; Adjustment for baseline
Statistical Analysis 6: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Ocular Surface Disease-Quality if Life (OSD-QoL®) dimension: Fear for the Future; Test type: Superiority; p = 0.0536, ANCOVA — Significance level of 0.05; Adjustment for baseline
Statistical Analysis 7: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Ocular Surface Disease-Quality if Life (OSD-QoL®) dimension: Emotional well-being; Test type: Superiority; p = 0.1998, ANCOVA — Significance level of 0.05; Adjustment for baseline
Statistical Analysis 8: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Ocular Surface Disease-Quality of Life (OSD-QoL®) questions: Global Question; Test type: Superiority; p = 0.0306, ANCOVA — Significance level of 0.05; Adjustment for baseline

8. Secondary Outcome: Change From Baseline in Tear Film Break Up Time (TFBUT) at Day 28 (Visit 4) and at Day 90 (Visit 5)
Description: The Tear Film Break Up Time (TFBUT) after fluorescein instillation, measured the time between the last blink and the first appearance of a dry spot or disruption of the tear film. The TFBUT was measured in tenth of seconds with a stopwatch provided to the sites. It was conducted 3 times and the means was calculated.
Time Frame: Baseline (Day 0), Visit 4 (Day 28), Visit 5 (Day 90)
Population: Per-protocol population. Two participants of the per-protocol population, one in each group, withdrew before the Day 90 (Visit 5).
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | CBL-102 Eye Drops | Vismed Multi Eye Drops
Number analyzed (Participants) | 45 | 34
seconds
  Change From Baseline Tear Film Break Up Time (TFBUT) at day 28 (Visit 4) | 1.2 (0.3) | 0.8 (0.3)
  Change From Baseline in Tear Film Break Up Time (TFBUT) at Day 90 (Visit 5): number analyzed (Participants) | 44 | 33
  Change From Baseline in Tear Film Break Up Time (TFBUT) at Day 90 (Visit 5) | 1.3 (0.2) | 0.7 (0.3)
Statistical Analysis 1: Comparison: CBL-102 Eye Drops vs Vismed Multi Eye Drops; Test type: Superiority; p > 0.05, ANCOVA — Significance level of 0.05; Adjustment for baseline

9. Secondary Outcome: Change From Baseline in Schirmer Test at Day 28 (Visit 4)
Description: Tear fluid secretion was assessed by the un-anaesthetized Schirmer test in the study eye with graduated strips in millimeters.
  Schirmer paper test strips were carefully inserted over the lower eyelid margin. The strips were removed after 5 minutes and the amount of tear fluid secretion ready to the nearest mm from the graduated strip margins.
Time Frame: Baseline (Day 0), Visit 4 (Day 28)
Population: Per -protocol population
Measure: Least Squares Mean (Standard Error); unit: mm/5 min
Arm/Group | CBL-102 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 45 | 34
mm/5 min | 1.2 (0.4) | 0.7 (0.5)
Statistical Analysis 1: Comparison: CBL-102 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p > 0.05, ANCOVA — Significance level 0.05; Adjustment for baseline

10. Secondary Outcome: Frequency of Eye Drop Instillation
Description: Mean daily frequency of investigational eye drop instillations as reported in participant's diary
Time Frame: From Day 0 to Day 90, an average of 3 months
Population: Two participants of the per-protocol population, one in each group withdrew before the Day 90 (Visit 5).
Measure: Mean (Standard Deviation); unit: drops per day
Arm/Group | CBL-102 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 44 | 33
drops per day | 3.4 (0.6) | 4.0 (1.0)
Statistical Analysis 1: Comparison: CBL-102 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p = 0.0017, Wilcoxon (Mann-Whitney) — Significance level of 0.05

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the whole treatment period from the first instillation until the last study visit (90 ± 10 days).
Description: Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not related to the investigational medical device. Adverse event reports were elicited from the participants or resulted from the assessments at each study visit and recorded
Groups:
- CBL-102 Eye Drops: Participants received CBL-102 Eye Drops, 3 to 6 times daily for 3 months in both eyes.
  CBL-102 Eye Drops: CE-marked medical device, tear substitute with 0.24% sodium hyaluronate, carbomer and triglycerides
  Safety population
- Vismed® Multi Eye Drops: Participants received Vismed® Multi eye drops, 3 to 6 times daily for 3 months in both eyes.
  Vismed® Multi: CE-marked medical device, tear substitute with 0.18% sodium hyaluronate
  Safety population
Arm/Group | CBL-102 Eye Drops | Vismed® Multi Eye Drops
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/47 | 0/39
Other Adverse Events (participants affected / at risk) | 0/47 | 2/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBL-102 Eye Drops (N=47) | Vismed® Multi Eye Drops (N=39)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — 76-year-woman was diagnosed with breast cancer after Day 28 visit. Study product stopped, no final visit. Remission of breast cancer after surgery & radiotherapy. Event was assessed as unrelated to study product or study procedure by investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBL-102 Eye Drops (N=47) | Vismed® Multi Eye Drops (N=39)
Eye discharge (Eye disorders) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The participants were not masked to treatment as the compared products were provided in their original bottles to maintain their aseptic conditions but all the bottles were relabelled with no trade name. Labels and outer packaging were identical except for randomization number. Participants received sealed boxes and returned sealed boxes with instructions to keep the investigator masked.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor have at least 60 days to review any publication or presentation. The first release of results will involve all sites in this multicenter study.

DOCUMENTS (2):
  • Study Protocol (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT03368404/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT03368404/SAP_001.pdf